CLINICAL TRIAL: NCT00664664
Title: A Randomized, Double-blind, Placebo-controlled Subjective Study to Assess the Efficacy of APD125 in Patients With Primary Insomnia Characterized by Difficulty Maintaining Sleep
Brief Title: Subjective Study to Assess the Efficacy of APD125 in Patients With Sleep Maintenance Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APD125-007
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Primary Insomnia
Keywords: insomnia; sleep maintenance insomnia; sleep quality; non-restorative sleep; multiple awakenings
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): APD125 20 mg
  Interventions: Drug: APD125
- 2 (Experimental): APD125 40 mg
  Interventions: Drug: APD125
- 3 (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD125 — soft gelatin capsule, 20 mg, daily dosing for up to 3 weeks
  Arms: 1
Drug: APD125 — soft gelatin capsule, 40 mg, daily dosing for up to 3 weeks
  Arms: 2
Drug: Placebo — soft gelatin capsule, daily dosing for up to 3 weeks
  Arms: 3

SUMMARY:
This study is designed to compare 2 doses of APD125 (20 mg and 40 mg) with placebo in otherwise healthy adults with primary insomnia primarily with complaints of maintaining sleep. Participants will be required to maintain a daily sleep dairy for up to 3 weeks while on study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 65 years
* Primary insomnia as defined in DSM-IV-TR, with predominant complaint of impaired sleep maintenance and confirmed by patient reported sleep diaries
* Generally good health

Exclusion Criteria:

* History of any sleep disorder, other than primary insomnia (e.g., restless leg syndrome, narcolepsy, sleep apnea, and disorders of REM/NREM sleep)
* Any clinically significant medical condition, laboratory finding, or ECG finding
* Pregnant and/or lactating females
* History of substance abuse within 2 years or positive urine drug screen
* Positive Hepatitis B/C results or HIV markers
* History of treatment with an investigational drug within the last month
* Recent travel involving crossing more than 3 time zones or plans to travel to another time zone (> 3 time zones) during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in subjective number of awakenings after sleep onset (sNAASO) | During and after 2 weeks of study drug

SECONDARY OUTCOMES:
Change from baseline in subjective total sleep time (sTST) | During and after 2 weeks on study drug
Change from baseline in subjective wake time after sleep onset (sWASO) | During and after 2 weeks on study drug
Change in subjective latency to sleep onset (sSLO) | During and after 2 weeks on study drug
Safety and tolerability as assessed by changes from baseline in adverse events, vital signs, 12-lead ECGs, physical examinations, and clinical laboratory values. | During and after 2 weeks on study drug

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (1):
- Arena Pharmaceuticals, Inc, San Diego, California, United States